CLINICAL TRIAL: NCT02814838
Title: A Phase 2, Multicentre, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of 400 mg Twice a Day Oral Ladarixin in Patients With New-onset Type 1 Diabetes
Brief Title: A Phase 2, Multicentre, Randomized, Double-blind, Placebo-controlled Study in Patients With New-onset Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEX0114; 2014-003968-20 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-06-28 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: Diabetes mellitus Type 1; Beta cells function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ladarixin (Experimental): Ladarixin oral capsule
  Interventions: Drug: Ladarixin
- Placebo (Placebo Comparator): Placebo oral capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ladarixin — Ladarixin oral capsule
  Other Names: Active treatment
  Arms: Ladarixin
Drug: Placebo — Placebo oral capsule
  Other Names: Placebo treatment
  Arms: Placebo

SUMMARY:
The objective of this clinical trial is to investigate whether ladarixin has sufficient activity (preservation of β-cell function and slow-down of the progression of T1D) to warrant its further development (proof of concept trial). The safety of ladarixin in the specific clinical setting will be also evaluated.

The study is a phase 2, multicentre, double-blind study. 72 patients with new-onset type 1 diabetes (T1D) were planned to be involved, randomly (2:1) assigned to receive either ladarixin treatment (400 mg b.i.d. for 3 cycles of 14 days on/14 days off - treatment group) or placebo (control group).

Recruitment was competitive among the study sites, until the planned number of patients was enrolled. A total of 76 patients were actually recruited.

DETAILED DESCRIPTION:
T1D is an organ-specific autoimmune disease in which the immune system attacks the insulin-producing β-cells. The onset of the disease typically occurs before adulthood and seriously affects a person's quality of life.

T1D is treated with life-long daily exogenous insulin injections and monitoring of blood glucose levels. However, even optimization of glucose control through the most recent technologies cannot adequately substitute for the finely tuned normal balance of the glucose levels. Therefore, despite marked improvements in diabetes care in recent years, insulin-dependent diabetes results in secondary long-term complications and is one of the leading causes of end-stage renal disease, blindness and amputation. Additionally, hypoglycaemia unawareness is a serious consequence of recurrent hypoglycaemia often requiring emergency care.

Maintenance of residual β-cell function (as measured by C-peptide response) was demonstrated to be associated with reduced rate of microvascular complications and hypoglycaemia, improved quality of life, and overall reduction in morbidity and associated management costs. Therefore, pharmacological approaches aimed at controlling the autoimmune response and restoring self-tolerance to pancreatic β-cells had attracted the clinical/scientific interest.

Among these, rituximab, CD3-specific monoclonal antibodies, GAD65, DiaPep277 have progressed to phase III clinical trials. Other agents, including cytokines modulators such as anti-TNF or anti-IL1, are under clinical evaluation. Unfortunately, even if safe preservation of β-cell function and improvement of glycaemic control have been evidenced for some of the pharmacological approaches evaluated so far, none has been definitely approved for the "treatment" of diabetes onset. New strategies are being evaluated which combine agents targeting sequential arms of the immune and inflammatory response involved in β-cell disruption. In this regard, IL-8 appears to be an important mediator in the progression of type 1 diabetes. Production and secretion of pro-inflammatory IL-8 has been demonstrated from human pancreatic islets upon enterovirus infections, and LPS-induced production of IL-8 by neutrophils is increased in type 1 pre-diabetic and diabetic patients. In parallel, circulating levels of IL-8 were elevated in children with T1D compared to non-diabetic controls. Specifically, levels of IL-8 correlate with glycaemic control, higher level being associated to poorer or unfavorable glucose control.

As a result of these findings, the modulation or inhibition of IL8 activity is considered a valid target for the development of innovative treatments aimed to control the progression of T1D.

Results obtained with ladarixin in mouse models of T1D, and particularly reversal of "diabetes" in the NOD mice, clearly showed the ability of this CXCR1/2 inhibitor to protect β-cells and either prevent or delay the progression of hyperglycaemia. The positive effects of ladarixin, coupled with the safety shown in phase 1 studies, provided a sound rationale for a clinical study aimed at evaluating the effect of ladarixin in patients with new onset diabetes and supported the conduct of the present study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18-45 years, inclusive;
2. New-onset T1D (randomization within 100 days from 1st insulin administration);
3. Positive for at least one diabetes-related auto-antibody (anti-GAD; IAA, if obtained within 10 days of the onset of insulin therapy; IA-2 antibody; ZnT8);
4. Require, or has required at some time, insulin, with the exclusion of patients taking twice daily pre-mixed insulin or on insulin pump;
5. Residual β-cell function as per peak stimulated (MMTT) C-peptide level >0.6ng/mL (0.2nmol/L); MMTT should not be performed within one week of resolution of a diabetic ketoacidosis event;
6. Patient able to comply with all protocol procedures for the duration of the study, including scheduled follow-up visits and examinations;
7. Patients who have given written informed consent prior of any study-related procedure not part of standard medical care.

Exclusion Criteria:

1. Patients taking twice daily pre-mixed insulin or on insulin pump;
2. Any other chronic disease, including type 2 diabetes, apart from autoimmune hypothyroidism requiring thyroid hormone replacement only; patients with severe (myxedema) disease potentially requiring immunosuppressive therapy will be excluded;
3. Moderate to severe renal impairment as per calculated creatinine clearance (CLcr) < 60 mL/min according to the Cockcroft-Gault formula (Cockcroft-Gault, 1976);
4. Hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L];
5. Hypoalbuminemia defined as serum albumin < 3 g/dL;
6. QTcF > 470 msec;
7. Complete Left Bundle Branch Block (LBBB), atrio-ventricular block (mobitz II 2nd degree or 2:1 atrio-ventricular block), complete heart block;
8. Electronic pacemaker positioned or implanted defibrillator;
9. History of significant cardiovascular disease;
10. Known hypersensitivity to non-steroidal antiinflammatory drugs;
11. Concomitant treatment with phenytoin, warfarin, sulphanylurea hypoglycemics (e.g. tolbutamide, glipizide, glibenclamide/glyburide, glimepiride, nateglinide) and high dose of amitriptyline (> 50 mg/day);
12. Previous (within 2 weeks prior to randomization) and concomitant treatment with metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors or amylin, or any medications known to influence glucose tolerance (e.g. β-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine antimalarial drugs, lithium, niacin, etc.);
13. Past (within 1 month prior to randomization) or current administration of any immunosuppressive medications (including oral, inhaled or systemically injected steroids) and use of any investigational agents, including any agents that impact the immune response or the cytokine system;
14. Pregnant or breast feeding women. Unwillingness to use effective contraceptive measures up to 2 months after the end of study drug administration (females and males). Effective contraceptive measures include an hormonal birth control (e.g. oral pills, long term injections, vaginal ring, patch); the intrauterine device (IUD); a double barrier method (e.g. condom or diaphragm plus spermicide foam).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, MD, Principal Investigator — Internal Medicine - Diabetes & Endocrinology Unit, San Raffaele Hospital Milan
Locations (8):
- Belgium (2):
  - Universitair Ziekenhuis Brussel Diabetes Clinic, Brussels
  - Universitair Ziekenhuis Leuven Campus Gasthuisberg Endocrinology, Leuven
- Germany (2):
  - Med. Klinik und Poliklinik 3, Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Zentrum für Diabetes und Gefäßerkrankungen, Münster
- Italy (4):
  - Università Aldo Moro-Ospedale Policlinico, Bari
  - Presidio Policlinico di Monserrato, Cagliari
  - Internal Medicine - Diabetes & Endocrinology Unit, San Raffaele Hospital Milan, Milan
  - Unità Operativa Complessa di Endocrinologia e Dialettologia. Università Campus Bio-Medico di Roma, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sordi V, Monti P, Lampasona V, Melzi R, Pellegrini S, Keymeulen B, Gillard P, Linn T, Bosi E, Rose L, Pozzilli P, Giorgino F, Cossu E, Piemonti L. Post hoc analysis of a randomized, double-blind, prospective trial evaluating a CXCR1/2 inhibitor in new-onset type 1 diabetes: endo-metabolic features at baseline identify a subgroup of responders. Front Endocrinol (Lausanne). 2023 Jun 20;14:1175640. doi: 10.3389/fendo.2023.1175640. eCollection 2023. PMID 37409229

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ladarixin | Placebo
Started | 50 | 26
Completed | 48 | 25
Not Completed | 2 | 1
Not completed — 3 agreed dates for the final visit missed | 1 | 0
Not completed — Consent withdrawal | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ladarixin | Placebo | Total
Number analyzed (Participants) | 50 | 26 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 26 | 76
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 29 | 16 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 49 | 26 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 20 | 11 | 31
  Italy | 17 | 10 | 27
  Germany | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC)(0-2 h) of C-peptide Response to the Mixed Meal Tolerance Test (MMTT) at Week 13
Description: C-peptide level is a widely used measure of pancreatic beta-cell function. The MMTT is one of the methods for its estimation. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each follow-up visit on weeks 13±1, 26±2, and 52±2.
  Prior to the test, patients withheld long-acting insulin on the morning of the test. Rapid-acting and short-acting insulin were allowed up to 6hrs and 2 hrs, respectively, before the test. The test was rescheduled if the patient had a capillary glucose value of >200mg/dL or <70mg/dL.
  After 2 pre-meal basal samples had been drawn between -20 to 0 min (basal 1 and basal 2), patients were given 6mL/kg of Boost® High Protein Nutritional Drink up to a maximum of 360mL, to be drunk within 5 min. Post-meal samples were drawn at 15, 30, 60, 90, 120 min after the meal at week 13+/-1 The 2-hour C-peptide AUC after the MMTT at Week 13±1 was transformed as log(x+1) values.
Time Frame: week 13±1
Population: ITT population: all patients who were randomised and received at least 1 dose of study treatment (either ladarixin or placebo)
Measure: Mean (Standard Deviation); unit: log(ng*hr/ml [0-2 h]+1)
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 49 | 26
log(ng*hr/ml [0-2 h]+1) | 4.026 (0.4852) | 3.886 (0.7446)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Transformed AUC was analyzed with Student t-test for unpaired data using PROC TTEST within SAS® to compare Ladarixin and placebo groups. The estimated treatment difference between Ladarixin and placebo was also presented together with the corresponding 95% confidence interval; Test type: Superiority; p = 0.3303, Student's t test for unpaired samples; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.14 to 0.42]

2. Secondary Outcome: Area Under the Curve (AUC) (0-2 h) of C-peptide Response to the Mixed Meal Tolerance Test (MMTT) at Weeks 26 and 52
Description: C-peptide level is a widely used measure of pancreatic beta-cell function. The MMTT is one of the methods for its estimation. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each follow-up visit on weeks 13±1, 26±2, and 52±2.
  Prior to the test, patients withheld long-acting insulin on the morning of the test. Rapid-acting and short-acting insulin were allowed up to 6hrs and 2 hrs, respectively, before the test. The test was rescheduled if the patient had a capillary glucose value of >200mg/dL or <70mg/dL. After 2 pre-meal basal samples had been drawn between -20 to 0 min (basal 1 and basal 2), patients were given 6mL/kg of Boost® High Protein Nutritional Drink up to a maximum of 360mL, to be drunk within 5 min. Post-meal samples were drawn at 15, 30, 60, 90, 120 min after the meal at week 13+/-1.
  The 2-hour C-peptide AUC after the MMTT at Week 13±1 was transformed as log(x+1) values.
Time Frame: Follow-ups at Weeks 26±2 and 52±2
Population: ITT population: all patients who were randomised and received at least 1 dose of study treatment (either ladarixin or placebo).
  Please note that the number of participants analysed represents the number of patients contributing to summary statistics.
Measure: Mean (Standard Deviation); unit: log(ng*hr/ml [0-2 h]+1)
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 47 | 25
log(ng*hr/ml [0-2 h]+1)
  FU week 26 | 3.9351 (0.51710) | 3.8076 (0.76473)
  FU week 52: number analyzed (Participants) | 46 | 25
  FU week 52 | 3.6371 (0.75222) | 3.6380 (0.81268)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at FUP week 26; Test type: Superiority — The comparisons between groups on 2-hour AUC C-peptide efficacy endpoint was carried-out using a mixed linear model where the log(x+1) transformed 2-hour AUC C-peptide was the dependent variable, while treatment group, visit, treatment by visit interaction were the fixed factors of the model and patient will be the random effect. An unstructured covariance matrix for each patient is considered and the Kenward-Roger adjustment is used for the degrees of freedom; p = 0.517, Mixed Models Analysis; adjusted mean difference = 0.0984, 95% CI 2-sided [-0.2028 to 0.3995]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At FUP week 52; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.7999, Mixed Models Analysis; adjusted mean difference = -0.0486, 95% CI 2-sided [-0.4294 to 0.3322]

3. Secondary Outcome: Percent Change From Baseline of 2-hour AUC of C-peptide Response to the MMTT
Description: C-peptide level is a widely used measure of pancreatic beta-cell function. The MMTT is one of the methods for its estimation. The MMTT was performed after an overnight fast, at baseline (within 1 week prior to randomization), and at each follow-up visit on weeks 13±1, 26±2, and 52±2.
  Prior to the test, patients withheld long-acting insulin on the morning of the test. Rapid-acting and short-acting insulin were allowed up to 6hrs and 2 hrs, respectively, before the test. The test was rescheduled if the patient had a capillary glucose value of >200mg/dL or <70mg/dL.
  The test was initiated before 10 a.m. After 2 pre-meal basal samples had been drawn between -20 to 0 min (basal 1 and basal 2), patients were given 6mL/kg of Boost® High Protein Nutritional Drink (Nestlé Nutrition) up to a maximum of 360mL, to be drunk within 5 min. Post-meal samples were drawn at 15±5, 30±5, 60±10, 90±10, 120±15, 180±15 min after the meal.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: ITT population = all patients who were randomised and received at least 1 dose of study treatment (either ladarixin or placebo).
  Please note that the number of participants analysed represents the number of patients contributing to summary statistics.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 49 | 25
percentage of change
  FU week 13 | 5.7818 (36.74477) | -6.0734 (38.22179)
  FU week 26: number analyzed (Participants) | 47 | 24
  FU week 26 | -0.8701 (42.93044) | -13.7347 (37.41900)
  FU week 52: number analyzed (Participants) | 46 | 24
  FU week 52 | -22.2532 (38.84672) | -24.2215 (42.67277)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority; p = 0.2224, Mixed Models Analysis; adjusted mean difference = 12.0411, 95% CI 2-sided [-7.3823 to 31.4644]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority; p = 0.3931, Mixed Models Analysis; adjusted mean difference = 8.4803, 95% CI 2-sided [-11.0935 to 28.0541]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At week 52; Test type: Superiority; p = 0.7664, Mixed Models Analysis; adjusted mean difference = -2.9502, 95% CI 2-sided [-22.5476 to 16.6473]

4. Secondary Outcome: Change From Screening in Average (Previous 3 Days) Insulin Requirement
Description: Insulin requirement (IU/kg/day averaged over the previous 3 days) was to be recorded in the interval from randomization to Week 13±1, Week 13±1 to Week 26±2, and Week 26±2 to Week 52±2.
  From enrolment, patients were admitted to intensive diabetes management, according to current ADA recommendation [2014]. Patients were instructed to self-monitor their glucose values at least 4 times a day and to report (glucose meter/log) outcome to the diabetes management team. Insulin intake was adjusted to target HbA1c levels of less than 7% and self-monitored (fingerstick):
  * pre-prandial blood glucose of 70-130 mg/dL
  * post-prandial blood glucose < 180 mg/dL
  * bed-time blood glucose of 110-150 mg/dL Telephone calls (outside scheduled visits) were scheduled on a regular basis to ensure optimization of metabolic control.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/kg/day
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 47 | 26
IU/kg/day
  FU week 13 | -0.067 (0.1774) | -0.018 (0.1314)
  FU week 26: number analyzed (Participants) | 47 | 25
  FU week 26 | -0.011 (0.2625) | 0.032 (0.1699)
  FU week 52: number analyzed (Participants) | 46 | 25
  FU week 52 | 0.025 (0.2507) | 0.101 (0.2411)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority — Analysis is based on a linear mixed model for repeated measures with Daily Insulin Requirement (IU/kg/day) as dependent variable, treatment, visit and treatment by visit interaction as fixed effects and patient as random effect; p = 0.2225, Mixed Models Analysis; adjusted mean difference = -0.048, 95% CI 2-sided [-0.1257 to 0.0298]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; at week 26; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.551, Mixed Models Analysis; adjusted mean difference = -0.0369, 95% CI 2-sided [-0.1596 to 0.0858]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; at week 52; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.2501, Mixed Models Analysis; adjusted mean difference = -0.063, 95% CI 2-sided [-0.1712 to 0.0453]

5. Secondary Outcome: Change From Screening in Glycated Haemoglobin (HbA1c) Levels
Description: HbA1c measurement can be used as a diagnostic test for diabetes providing that stringent quality assurance tests are in place and assays are standardised to criteria aligned to the international reference values, and there are no conditions present which preclude its accurate measurement.
  An HbA1c of 6.5% is recommended as the cut point for diagnosing diabetes. A value of less than 6.5% does not exclude diabetes diagnosed using glucose tests.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 48 | 25
percentage of glycated haemoglobin
  FU week 13 | -1.40 (1.674) | -1.18 (1.352)
  FU week 26: number analyzed (Participants) | 47 | 24
  FU week 26 | -1.19 (2.003) | -0.63 (1.141)
  FU week 52: number analyzed (Participants) | 46 | 25
  FU week 52 | -0.69 (2.225) | -0.76 (1.333)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at FU week 13; Test type: Superiority — Analysis is based on a linear mixed model for repeated measures with HbA1c (%) as dependent variable, treatment, visit and treatment by visit interaction as fixed effects and patient as random effect; p = 0.6252, Mixed Models Analysis; adjusted mean difference = -0.1494, 95% CI 2-sided [-0.7514 to 0.4526]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At FU week 26; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.366, Mixed Models Analysis; adjusted mean difference = -0.2804, 95% CI 2-sided [-0.8904 to 0.3297]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At FU week 52; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.5026, Mixed Models Analysis; adjusted mean difference = -0.2063, 95% CI 2-sided [-0.3992 to 0.8118]

6. Secondary Outcome: Basal to 180 Minutes Time Course of C-peptide Concentration Derived From the MMTT
Description: Time points at each visit are Basal 1 and Basal 2 (samples collected at -20 and 0 min, respectively; Here are reported the following timepoints: Basal average (which is the average of Basal 1 and Basal 2), 15, 30, 60, 90, 120, and 180 minutes after the meal. For values at each time point see below.
Time Frame: Baseline, follow-ups at Weeks 13±1, 26±2, and 52±2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 50 | 26
nmol/L
  Screening - Basal average | 0.218 (0.1087) | 0.225 (0.1416)
  Screening - 15 min | 0.294 (0.1621) | 0.299 (0.1779)
  Screening - 30 min | 0.422 (0.2126) | 0.452 (0.3036)
  Screening - 60 min: number analyzed (Participants) | 50 | 25
  Screening - 60 min | 0.545 (0.2631) | 0.537 (0.2354)
  Screening - 90 min: number analyzed (Participants) | 50 | 25
  Screening - 90 min | 0.613 (0.2467) | 0.581 (0.2486)
  Screening - 120 min: number analyzed (Participants) | 49 | 26
  Screening - 120 min | 0.620 (0.2559) | 0.656 (0.2923)
  Screening - 180 min: number analyzed (Participants) | 49 | 25
  Screening - 180 min | 0.527 (0.2252) | 0.550 (0.2277)
  week 13 - Basal average: number analyzed (Participants) | 49 | 26
  week 13 - Basal average | 0.231 (0.1136) | 0.210 (0.1315)
  week 13 - 15 min: number analyzed (Participants) | 49 | 26
  week 13 - 15 min | 0.300 (0.1385) | 0.285 (0.1956)
  week 13 - 30 min: number analyzed (Participants) | 49 | 26
  week 13 - 30 min | 0.427 (0.2048) | 0.392 (0.2418)
  week 13 - 60 min: number analyzed (Participants) | 49 | 26
  week 13 - 60 min | 0.571 (0.2660) | 0.523 (0.2729)
  week 13 - 90 min: number analyzed (Participants) | 49 | 26
  week 13 - 90 min | 0.620 (0.2859) | 0.594 (0.3176)
  week 13 - 120 min: number analyzed (Participants) | 49 | 26
  week 13 - 120 min | 0.637 (0.2869) | 0.601 (0.3050)
  week 13 - 180 min: number analyzed (Participants) | 48 | 26
  week 13 - 180 min | 0.518 (0.2302) | 0.527 (0.2778)
  week 26 - Basal average: number analyzed (Participants) | 47 | 25
  week 26 - Basal average | 0.212 (0.0941) | 0.207 (0.1192)
  week 26 - 15 min: number analyzed (Participants) | 47 | 25
  week 26 - 15 min | 0.278 (0.1294) | 0.260 (0.1426)
  week 26 - 30 min: number analyzed (Participants) | 47 | 25
  week 26 - 30 min | 0.391 (0.1857) | 0.368 (0.2150)
  week 26 - 60 min: number analyzed (Participants) | 47 | 25
  week 26 - 60 min | 0.534 (0.2463) | 0.511 (0.2967)
  week 26 - 90 min: number analyzed (Participants) | 47 | 25
  week 26 - 90 min | 0.569 (0.2606) | 0.552 (0.3101)
  week 26 - 120 min: number analyzed (Participants) | 46 | 25
  week 26 - 120 min | 0.592 (0.2703) | 0.552 (0.2907)
  week 26 - 180 min: number analyzed (Participants) | 47 | 25
  week 26 - 180 min | 0.504 (0.2189) | 0.466 (0.2362)
  week 52 - Basal average: number analyzed (Participants) | 46 | 25
  week 52 - Basal average | 0.168 (0.1070) | 0.178 (0.1068)
  week 52 - 15 min: number analyzed (Participants) | 46 | 25
  week 52 - 15 min | 0.228 (0.1606) | 0.249 (0.1616)
  week 52 - 30 min: number analyzed (Participants) | 46 | 25
  week 52 - 30 min | 0.321 (0.2231) | 0.314 (0.1826)
  week 52 - 60 min: number analyzed (Participants) | 46 | 25
  week 52 - 60 min | 0.430 (0.2693) | 0.440 (0.2671)
  week 52 - 90 min: number analyzed (Participants) | 46 | 25
  week 52 - 90 min | 0.463 (0.2806) | 0.465 (0.2881)
  week 52 - 120 min: number analyzed (Participants) | 46 | 25
  week 52 - 120 min | 0.503 (0.3085) | 0.492 (0.2717)
  week 52 - 180 min: number analyzed (Participants) | 46 | 25
  week 52 - 180 min | 0.426 (0.2341) | 0.443 (0.2441)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority — Analysis is based on a linear mixed model for repeated measures with C-peptide (nmol/L) actual value as dependent variable, treatment, visit, time, treatment by visit interaction, time by visit interaction, treatment by visit by time interaction as fixed effects and time by visit interaction is specified in repeated statement; p = 0.2527, Mixed Models Analysis; adjusted mean difference = 0.0242, 95% CI 2-sided [-0.0174 to 0.0658]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; at week 26; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.2743, Mixed Models Analysis; adjusted mean difference = 0.0236, 95% CI 2-sided [-0.0188 to 0.066]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; at week 52; Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.7856, Mixed Models Analysis; adjusted mean difference = -0.0059, 95% CI 2-sided [-0.0485 to 0.0367]

7. Secondary Outcome: Basal to 180 Minutes Time Course of Glucose Concentration Derived From the MMTT
Description: Time points at each visit are Basal 1 and Basal 2 (samples collected at -20 and 0 min, respectively). Here are reported the following timepoints: Basal average (which is the average of Basal 1 and Basal 2), 15, 30, 60, 90, 120, and 180 minutes after the meal. For values at each time point see below.
Time Frame: Baseline, follow-ups at Weeks 13±1, 26±2, and 52±2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 50 | 26
mmol/L
  Screening - basal average | 6.965 (1.6858) | 6.855 (1.9507)
  Screening - 15 min | 8.108 (1.8453) | 8.013 (2.0941)
  Screening - 30 min | 10.438 (2.2282) | 10.096 (2.4694)
  Screening - 60 min: number analyzed (Participants) | 50 | 25
  Screening - 60 min | 12.146 (2.9387) | 12.068 (2.9204)
  Screening - 90 min: number analyzed (Participants) | 50 | 25
  Screening - 90 min | 12.350 (3.4122) | 12.076 (3.9156)
  Screening - 120 min | 11.400 (3.4561) | 11.827 (4.0204)
  Screening - 180 min: number analyzed (Participants) | 49 | 25
  Screening - 180 min | 9.478 (3.6320) | 9.652 (4.0549)
  Week 13 - Basal average: number analyzed (Participants) | 49 | 25
  Week 13 - Basal average | 7.074 (1.9973) | 6.644 (2.1145)
  Week 13 - 15 min: number analyzed (Participants) | 49 | 25
  Week 13 - 15 min | 8.231 (2.1415) | 7.836 (2.2409)
  Week 13 - 30 min: number analyzed (Participants) | 49 | 25
  Week 13 - 30 min | 10.727 (2.5691) | 10.224 (2.3600)
  Week 13 - 60 min: number analyzed (Participants) | 49 | 24
  Week 13 - 60 min | 12.614 (3.1536) | 12.871 (2.6908)
  Week 13 - 90 min: number analyzed (Participants) | 49 | 25
  Week 13 - 90 min | 12.553 (3.7998) | 13.092 (3.1608)
  Week 13 - 120 min: number analyzed (Participants) | 49 | 25
  Week 13 - 120 min | 11.773 (4.0990) | 12.260 (3.7590)
  Week 13 - 180 min: number analyzed (Participants) | 49 | 25
  Week 13 - 180 min | 9.761 (3.9834) | 9.984 (3.8597)
  Week 26 - Basal average: number analyzed (Participants) | 48 | 25
  Week 26 - Basal average | 7.496 (2.0261) | 7.600 (2.6387)
  Week 26 - 15 min: number analyzed (Participants) | 48 | 24
  Week 26 - 15 min | 8.750 (2.0827) | 9.058 (2.7026)
  Week 26 - 30 min: number analyzed (Participants) | 48 | 25
  Week 26 - 30 min | 10.927 (2.3901) | 11.240 (2.6187)
  Week 26 - 60 min: number analyzed (Participants) | 48 | 25
  Week 26 - 60 min | 13.494 (2.8623) | 14.222 (2.8795)
  Week 26 - 90 min: number analyzed (Participants) | 48 | 25
  Week 26 - 90 min | 13.665 (3.8399) | 15.020 (3.4469)
  Week 26 - 120 min: number analyzed (Participants) | 48 | 25
  Week 26 - 120 min | 13.240 (4.1302) | 14.424 (3.7761)
  Week 26 - 180 min: number analyzed (Participants) | 48 | 25
  Week 26 - 180 min | 10.956 (4.2031) | 12.028 (3.8832)
  Week 52 - Basal average: number analyzed (Participants) | 46 | 25
  Week 52 - Basal average | 7.457 (2.3045) | 8.163 (2.2251)
  Week 52 - 15 min: number analyzed (Participants) | 46 | 25
  Week 52 - 15 min | 8.939 (2.7210) | 9.544 (2.2230)
  Week 52 - 30 min: number analyzed (Participants) | 46 | 25
  Week 52 - 30 min | 11.374 (2.6806) | 11.688 (2.6411)
  Week 52 - 60 min: number analyzed (Participants) | 46 | 24
  Week 52 - 60 min | 14.315 (3.1205) | 14.725 (2.9631)
  Week 52 - 90 min: number analyzed (Participants) | 46 | 25
  Week 52 - 90 min | 14.911 (3.5768) | 15.276 (3.7144)
  Week 52 - 120 min: number analyzed (Participants) | 46 | 25
  Week 52 - 120 min | 14.354 (3.9162) | 15.140 (3.7514)
  Week 52 - 180 min: number analyzed (Participants) | 46 | 25
  Week 52 - 180 min | 12.148 (4.0817) | 13.148 (3.9136)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority — Analysis is based on a linear mixed model for repeated measures with Glucose (mmol/L) actual value as dependent variable, treatment, visit, time, treatment by visit interaction, time by visit interaction, treatment by visit by time interaction as fixed effects and time by visit interaction is specified in repeated statement; p = 0.9307, Mixed Models Analysis; adjusted mean difference = -0.0253, 95% CI 2-sided [-0.5986 to 0.548]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.0139, Mixed Models Analysis; adjusted mean difference = -0.7236, 95% CI 2-sided [-1.2989 to -0.1483]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; at week 52; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.0432, Mixed Models Analysis; adjusted mean difference = -0.5979, 95% CI 2-sided [-1.1775 to -0.0184]

8. Secondary Outcome: Cumulative Severe Hypoglycaemic Events Occurring From Randomisation by Visit
Description: A severe hypoglycaemic event was defined as an event with one of the following symptoms: "memory loss, confusion, uncontrollable behaviour, irrational behaviour, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the patient was unable to treat him/herself and which was associated with either a blood glucose level <54 mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 50 | 26
events
  FU week 13: number analyzed (Participants) | 49 | 26
  FU week 13 | 0.0 (0.0) | 0.0 (0.0)
  FU Week 26: number analyzed (Participants) | 48 | 25
  FU Week 26 | 0.0 (0.14) | 0.0 (0.20)
  FU Week 52: number analyzed (Participants) | 49 | 25
  FU Week 52 | 0.1 (0.32) | 0.0 (0.20)

9. Secondary Outcome: Proportion of Patients Maintaining a Residual β-cell Function
Description: Maintenance of a residual ß-cell function is defined as at least one MMTT C-peptide value > 0.2 nmol/L.
  Proportion is reported as Percentage of patients.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: ITT population = all patients who were randomised and received at least 1 dose of study treatment (either ladarixin or placebo)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 49 | 26
Percentage of patients
  FU Week 13 | 96.0 [86.29 to 99.51] | 88.5 [69.85 to 97.55]
  FU week 26: number analyzed (Participants) | 46 | 25
  FU week 26 | 86.0 [73.26 to 94.18] | 84.6 [65.13 to 95.64]
  FU Week 52: number analyzed (Participants) | 45 | 25
  FU Week 52 | 78.0 [64.04 to 88.47] | 76.9 [56.35 to 91.03]
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority; p = 0.1171, Fisher Exact
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority; p = 0.6586, Fisher Exact
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At week 52; Test type: Superiority; p = 0.5056, Fisher Exact

10. Secondary Outcome: Proportion of Patients With HbA1c <7% and Absence of Episodes of Severe Hypoglycaemia From the Previous Visit
Description: A severe hypoglycaemic event was defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behaviour, irrational behaviour, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the patient was unable to treat him/herself and which was associated with either a blood glucose level <54 mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
  Proportion is reported as percentage of patients. Events per patient are calculated from the date of randomisation.
Time Frame: Follow-ups at Weeks 13±1, 26±2 and 52±2
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 49 | 25
Percentage of patients
  FU Week 13 | 90.0 [78.19 to 96.67] | 73.1 [52.21 to 88.43]
  FU week 26: number analyzed (Participants) | 48 | 24
  FU week 26 | 78.0 [64.04 to 88.47] | 50.0 [29.93 to 70.07]
  FU Week 52: number analyzed (Participants) | 47 | 25
  FU Week 52 | 62.0 [47.17 to 75.35] | 53.8 [33.37 to 73.41]
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; at week 13; Test type: Superiority; p = 0.0779, Fisher Exact
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority; p = 0.0248, Fisher Exact
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At week 52; Test type: Superiority; p = 0.4504, Fisher Exact

11. Secondary Outcome: C-peptide AUC(15 to 120 Mins) Above Fasting Value
Description: The means are all "adjusted means". The MMTT over the study: logAUC(15-120 min) of C-peptide above fasting value at Weeks 13±1, 26±2, and 52±2 is reported.
  Post-meal samples were drawn at 15, 30, 60, 90, 120 min after the meal at weeks 13+/-1, 26±2 and 52±2
Time Frame: Follow-ups at Weeks 13±1 26±2 and 52±2
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: log(ng*hr/ml [15-120 min]+1)
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 50 | 26
log(ng*hr/ml [15-120 min]+1)
  FU Week 13 | 3.3736 [3.1730 to 3.5742] | 3.2334 [2.9568 to 3.5100]
  FU week 26 | 3.2419 [3.0186 to 3.4652] | 3.0649 [2.7562 to 3.3735]
  FU week 52 | 2.9733 [2.7150 to 3.2316] | 2.9282 [2.5720 to 3.2844]
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; At week 13; Test type: Superiority — Analysis is based on a linear mixed model for repeated measures with log(AUC(15-120 minutes)+1) of C-peptide above fasting value as dependent variable, treatment, visit and treatment by visit interaction as fixed effects and patient as random effect; p = 0.4163, Mixed Models Analysis; adjusted mean difference = 0.1402, 95% CI 2-sided [-0.2015 to 0.4819]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.3575, Mixed Models Analysis; adjusted mean difference = 0.177, 95% CI 2-sided [-0.2039 to 0.558]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At week 52; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.8386, Mixed Models Analysis; adjusted mean difference = 0.0451, 95% CI 2-sided [-0.3948 to 0.4851]

12. Secondary Outcome: Area Under the Curve (AUC) (0-2 h) of C-peptide MMTT in Patients With Screening C-peptide < Median Value
Description: A subgroup analysis of efficacy endpoints by fasting C-peptide at Screening was performed. The reported data specifically refers to fasting C-peptide at Screening <median value. All the AUC analyses were based on actual rather than scheduled timings and were calculated using the trapezoidal rule. If the actual time was not recorded, the scheduled time was used instead. Post-meal samples were drawn at 15, 30, 60, 90, 120 min after the meal.
  The 2-hour C-peptide AUC after the MMTT was transformed as log(x+1) values.
Time Frame: Follow-up at Weeks 13±1, 26±2, and 52±2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log(ng*hr/ml [0-2 h]+1)
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 26 | 11
log(ng*hr/ml [0-2 h]+1)
  FU Week 13 | 3.8085 (0.45692) | 3.4543 (0.86632)
  FU Week 26: number analyzed (Participants) | 25 | 10
  FU Week 26 | 3.8202 (0.48142) | 3.3178 (0.91906)
  FU Week 52: number analyzed (Participants) | 24 | 10
  FU Week 52 | 3.3796 (0.68616) | 3.1562 (0.97130)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; At week 13; Test type: Superiority — Transformed AUC was analyzed with Student t-test for unpaired data using PROC TTEST within SAS® to compare Ladarixin and placebo groups. The estimated treatment difference between Ladarixin and placebo was also presented together with the corresponding 95% confidence interval; p = 0.1114, t-test, 2 sided; Mean Difference (Final Values) = 0.354, 95% CI 2-sided [-0.09 to 0.75]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; At week 26; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.0411, t-test, 2 sided; Mean Difference (Final Values) = 0.502, 95% CI 2-sided [0.02 to 0.98]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; At week 52; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p = 0.4506, t-test, 2 sided; Mean Difference (Final Values) = 0.223, 95% CI 2-sided [-0.37 to 0.82]

13. Secondary Outcome: Area Under the Curve (AUC) (15-120 Min) of C-peptide MMTT Above Fasting Value in Patients With Screening C-peptide < Median Value
Description: A subgroup analysis of efficacy endpoints by fasting C-peptide at Screening was performed. The reported data specifically refers to fasting C-peptide at Screening <median value. All the AUC analyses were based on actual rather than scheduled timings and were calculated using the trapezoidal rule. If the actual time was not recorded, the scheduled time was used instead.
  Post-meal samples were drawn at 15, 30, 60, 90, 120 min after the meal at Weeks 13±1, 26±2, and 52±2.
Time Frame: Follow-up at Weeks 13±1, 26±2, and 52±2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: log(ng*hr/ml [15-120 min] +1)
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 26 | 11
log(ng*hr/ml [15-120 min] +1)
  FU week 13 | 3.1590 (0.56135) | 2.7959 (1.07745)
  FU week 26: number analyzed (Participants) | 25 | 10
  FU week 26 | 27.7841 (15.10337) | 18.6842 (15.46837)
  FU week 52: number analyzed (Participants) | 24 | 10
  FU week 52 | 2.7993 (0.82214) | 19.9415 (16.95597)
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Week 13 Analysis is based on a linear mixed model for repeated measures with log(AUC(15-120 minutes)+1) of C-peptide above fasting value as dependent variable, treatment, visit and treatment by visit interaction; Test type: Superiority; p = 0.1847, Mixed Models Analysis; Adjusted mean difference = 0.3631, 95% CI 2-sided [-0.1817 to 0.908]
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Week 26 Analysis is based on a linear mixed model for repeated measures with log(AUC(15-120 minutes)+1) of C-peptide above fasting value as dependent variable, treatment, visit and treatment by visit interaction; Test type: Superiority; p = 0.031, Mixed Models Analysis; Adjusted mean difference = 0.6304, 95% CI 2-sided [0.0609 to 1.1998]
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Week 52 Analysis is based on a linear mixed model for repeated measures with log(AUC(15-120 minutes)+1) of C-peptide above fasting value as dependent variable, treatment, visit and treatment by visit interaction; Test type: Superiority; p = 0.6299, Mixed Models Analysis; Adjusted mean difference = 0.1639, 95% CI 2-sided [-0.5202 to 0.8479]

14. Secondary Outcome: Proportion of Patients With HbA1c <7% and Absence of Episodes of Severe Hypoglycaemia From the Previous Visit in Patients With Screening C-peptide < Median Value
Description: A severe hypoglycaemic event was defined as an event with one of the following symptoms: memory loss, confusion, uncontrollable behaviour, irrational behaviour, unusual difficulty in awakening, suspected seizure, seizure, loss of consciousness, or visual symptoms", in which the patient was unable to treat him/herself and which was associated with either a blood glucose level <54 mg/dL or prompt recovery after oral carbohydrate, i.v. glucose, or glucagon administration.
  Proportion is reported as percentage of patients, despite the measure type indicated is "number".
  Events per patient are calculated from the date of randomisation.
Time Frame: Follow-up at Weeks 13±1, 26±2, and 52±2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Ladarixin | Placebo
Number analyzed (Participants) | 26 | 11
Percentage of patients
  FU week 13 | 88.5 [69.85 to 97.55] | 63.6 [30.79 to 89.07]
  FU week 26: number analyzed (Participants) | 25 | 9
  FU week 26 | 88.5 [69.85 to 97.55] | 36.4 [10.93 to 69.21]
  FU week 52: number analyzed (Participants) | 25 | 10
  FU week 52 | 65.4 [44.33 to 82.79] | 45.5 [16.75 to 76.62]
Statistical Analysis 1: Comparison: Ladarixin vs Placebo; Week 13; Test type: Superiority; p = 0.163, Fisher Exact
Statistical Analysis 2: Comparison: Ladarixin vs Placebo; Week 26; Test type: Superiority; p = 0.0074, Fisher Exact
Statistical Analysis 3: Comparison: Ladarixin vs Placebo; Week 52; Test type: Superiority; p = 0.4437, Fisher Exact

ADVERSE EVENTS:
Time Frame: AEs were recorded and reported in the CRF from enrollment throughout patient's participation in the study (last planned visit or early withdrawal date), an average of 3 years
Arm/Group | Ladarixin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/26
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/26
Other Adverse Events (participants affected / at risk) | 37/50 | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladarixin (N=50) | Placebo (N=26)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ladarixin (N=50) | Placebo (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (9) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gatroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (4)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 2 (3)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroeteritis viral (Infections and infestations) | 1 (1) | 3 (3)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (2)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 13 (19) | 4 (6)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Eosinophil count decreased (Investigations) | 0 (0) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (7) | 1 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 14 (20) | 6 (8)
Migrane (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional distress (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (4) | 0 (0)
Nipple inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Increased viscosity of upper respiratiory secretion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT02814838/Prot_001.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT02814838/SAP_000.pdf